CLINICAL TRIAL: NCT03268642
Title: Assesment of Clinical Therapeutic Efficacy of "Life-support Based Comprehensive Treatment Regimen" for Adult Fulminant Myocarditis
Brief Title: Clinical Assessment of New Treatment Regimen for Adult Fulminant Myocarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Principal Investigator, Tongji Hospital
Other Study IDs: TJH-C20160202
Record Dates: First submitted 2017-08-17; First posted 2017-08-31 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Fulminant Myocarditis
Keywords: Fulminant Myocarditis; Retrospective cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Life-support Based Comprehensive Treatment Regimen group: meet all the following conditions:
  1. intravenous immune globulin;
  2. large dose of glucocorticoids;
  3. mechanical ventilation;
  4. hemodynamic support: intra-aortic balloon pump (IABP) or/and extracorporeal membrane oxygenation (ECMO);
  5. continuous renal replacement therapy.
- conventional therapy group: meet one of the following conditions:
  1. without/insufficient intravenous immune globulin;
  2. without/with various doses of glucocorticoid ;
  3. vasoactive drug;
  4. without/delayed mechanical ventilation;
  5. without/delayed hemodynamic support;
  6. without/delayed continuous renal replacement therapy.

SUMMARY:
This is a retrospective cohort study to assess the clinical outcome of patients with fulminant myocarditis using "Life-support Based Comprehensive Treatment Regimen" and conventional therapy. In the present study, participants receive various treatment as part of routine medical care without any assignment of specific interventions to them. The process of treatment during hospitalization were recorded in medical chart and was reviewed by independent research personnel.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older;
* Diagnosed as fulminant myocarditis:

  * Evidence of myocarditis on biopsy or increased biomarkers of myocardial injury (TNI and CK-MB and BNP or NT-pro-BNP);
  * Acute onset of symptoms of cardiac dysfunction: dyspnea, palpation, chest pain, and/or syncope;
  * Image for cardiac injury: marked diffused reduction in left ventricle wall movement, with dramatically decreased left ventricle ejection fraction (LVEF) < 45%;
  * Cardiogenic shock, e.g., systolic blood pressure ≤90 mmHg or mean arterial pressure < 70mm Hg or a systolic blood pressure decrease > 40 mm Hg, which is associated with the signs of hypofusion: cyanosis, cold extremities, oliguria, and/or changes in mental status.

Exclusion Criteria:

* Also considering acute coronary syndrome but unable to perform coronary angiography to distinguish acute coronary syndrome from fulminant myocarditis;
* Myocardial injury caused by sepsis, chemotherapeutical agents, or poisons;
* Unstable hemodynamics or shock caused by hypovolemia.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 150 hospitalized patients with fulminant myocarditis will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-02-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
death or cardiac transplantation | through hospital discharge, an average of 10 days
  The occurrence of death or cardiac transplantation was determined through direct contact with the patient or the family of the patient or review of the patient's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Cui G, Nie J, Li H, Wang L, Miao K, Zhao C, Jiang J, Wang DW. The clinicopathologic features of fulminant myocarditis. J Adv Res. 2025 Jun 18:S2090-1232(25)00449-7. doi: 10.1016/j.jare.2025.06.040. Online ahead of print. PMID 40541779
- [Derived] He W, Wu J, Wang D, Chen W, Yan Y, He Q, Li C, Yang Q, Huang C, Wen Z, Chen C, He F, Tang L, Wang DW. Plasma proteomics identifies S100A8/A9 as a novel biomarker and therapeutic target for fulminant myocarditis. J Adv Res. 2025 Jun 4:S2090-1232(25)00391-1. doi: 10.1016/j.jare.2025.06.005. Online ahead of print. PMID 40480626
- [Derived] Wang J, He M, Li H, Chen Y, Nie X, Cai Y, Xie R, Li L, Chen P, Sun Y, Li C, Yu T, Zuo H, Cui G, Miao K, Zhao C, Jiang J, Heidecker B, Barnett O, Maisel A, Chen C, Wang DW. Soluble ST2 Is a Sensitive and Specific Biomarker for Fulminant Myocarditis. J Am Heart Assoc. 2022 Apr 5;11(7):e024417. doi: 10.1161/JAHA.121.024417. Epub 2022 Apr 4. PMID 35377184